CLINICAL TRIAL: NCT00753909
Title: Paclitaxel, Carboplatin Plus Bevacizumab in Pretreated, Advanced or Metastatic Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.17
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Paclitaxel; Carboplatin; Bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Bevacizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Paclitaxel/Carboplatin/Bevacizumab
  Interventions: Drug: Carboplatin; Drug: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Carboplatin (IV) 3 AUC on day 1 and day 15 every 4 weeks for 6 cycles
Drug: Bevacizumab — Bevacizumab (IV) 10 mg/kg on day 1 and day 15 every 4 weeks for 6 cycles Followed by Bevacizumab (IV) 15 mgr/Kgr on day 1 every 3 weeks until disease progression
  Other Names: Avastin
Drug: Paclitaxel — Paclitaxel (IV) 140 mg/m2,on day 1 and day 15 every 4 weeks for 6 cycles
  Other Names: Taxoprol; Paxene; Taxol

SUMMARY:
This trial will evaluate the efficacy and safety of paclitaxel, carboplatin and bevacizumab combination, administered biweekly, in patients with pretreated, advanced non small cell lung cancer.

DETAILED DESCRIPTION:
The addition of bevacizumab to paclitaxel plus carboplatin in the 1st line treatment of patients with advanced or metastatic non small cell lung cancer (NSCLC) provided a survival benefit. There are patients with NSCLC who have not received bevacizumab and have relapsed after 1st and/or 2nd line therapy. The evaluation of bevacizumab plus chemotherapy in such patients is justified. The combination of paclitaxel and carboplatin, administered every two weeks, has a favorable toxicity profile. This study will evaluate the addition of bevacizumab to a biweekly regimen of paclitaxel and carboplatin as 2nd or 3rd line therapy for NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, unresectable locally advanced (stage IIIB) or metastatic (stage IV) non-squamous NSCLC
* Non-squamous histologic type
* At least one and no more than two previous chemotherapy regimens for advanced or metastatic NSCLC
* Measurable disease, defined as at least 1 bidimensionally measurable lesion ≥ 20 X 10 mm.
* Age ≥ 18 years
* Performance status (WHO) 0-2
* Life expectancy of at least 12 weeks
* Adequate bone marrow (ANC ≥ 1,500/mm3, PLT ≥ 100,000/mm3, Hgb ≥ 9 g/dL), liver (Bilirubin ≤ 1.5 upper normal limit, SGOT/SGPT ≤ 2.5 upper normal limit in the absence of liver metastases or ≤ 5 upper normal limit in the presence of liver metastases), and renal function (Creatinine ≤ 1,5 upper normal limit)
* Patients must be able to understand the nature of this study
* Written informed consent

Exclusion Criteria:

* Previous therapy with paclitaxel in combination with carboplatin
* Second primary malignancy, except for non-melanoma skin cancer and in situ cervical cancer
* Pregnant or lactating women
* Any serious, uncontrolled comorbidity on the investigator's judgment
* Uncontrolled infection
* Any sustained chronic toxicity > grade 2 according to the NCI CTCAE (version 3.0)
* Symptomatic neuropathy > grade 2 according to the NCI CTCAE (version 3.0)
* Brain metastases, except if radiated and asymptomatic
* Radiotherapy within the previous 4 weeks
* Previous radiotherapy to the only measurable lesion
* Proteinuria ≥ 500 mgr of protein daily
* Hemoptysis > 10 cc per event
* Clinically significant hematemesis
* Centrally located lesion or in contact with major vessels
* Pulmonary lesion with cavitation
* Documented hemorrhagic diathesis or coagulation disorder
* Cardiovascular disease (class II-IV NYHA congestive heart failure, myocardial infarction within the previous 4 months, unstable angina, LVEF < normal, ventricular arrhythmia, uncontrolled hypertension)
* Thrombotic event within the previous 6 months
* Concurrent use of aspirin > 325 mgr daily, low molecular weight heparin in therapeutic dose, warfarin or acenocoumarol, non-steroid anti-inflammatory agents
* Concurrent treatment with other anti-cancer drug
* Major surgical procedure within the previous 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)

SECONDARY OUTCOMES:
Toxicity profile | Toxicity assessment of each chemotherapy cycle
Time to Tumor Progression | 1-year
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Agelaki, MD, Principal Investigator — University Hospital of Crete
Locations (10):
- Greece (10):
  - University Hospital of Heraklion, Dep of Medical Oncology, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Diabalkaniko" hospital, Thessaloniki, Thessaloniki
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki